CLINICAL TRIAL: NCT03612388
Title: Combined Use of a Novel Cardioplegic Formula With MPS® Versus Cardioplexol ® in Isolated CABG Using MiECC (Minimal Extracorporeal Circulation System)
Brief Title: Combined Use of a Novel Cardioplegic Formula With Myocardial Protection System (MPS)® Versus Cardioplexol ® in Isolated Coronary Artery Bypass Grafting (CABG) Using MiECC;
Acronym: MiECC
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00926; ch18Reuthebuch3
Record Dates: First submitted 2018-07-17; First posted 2018-08-02 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Complication of Extracorporeal Circulation; Complication of Coronary Artery Bypass Graft
MeSH Terms: interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cardioplegia with MPS® (Myocardial protection system): cardioplegic formula with MPS® (Myocardial protection system); use of a cardioplegic formula in isolated CABG (coronary artery bypass grafting) using MiECC (Minimal extracorporeal circulation
  Interventions: Procedure: use of a cardioplegic formula in isolated CABG (coronary artery bypass grafting) using MiECC (Minimal extracorporeal circulation
- cardioplegia with Cardioplexol ®: cardioplegic formula with Cardioplexol ® (colloid solution with Procaine, magnesium and potassium)

INTERVENTIONS:
Procedure: use of a cardioplegic formula in isolated CABG (coronary artery bypass grafting) using MiECC (Minimal extracorporeal circulation — use of a novel cardioplegic formula with MPS® (Myocardial protection system) versus Cardioplexol ® (colloid solution with Procaine, magnesium and potassium) in isolated CABG (coronary artery bypass grafting) using MiECC (Minimal extracorporeal circulation system).
  Groups: cardioplegia with MPS® (Myocardial protection system)

SUMMARY:
Combined use of a novel cardioplegic formula with MPS® (Myocardial protection system) versus Cardioplexol ® (colloid solution with Procaine, magnesium and potassium) in isolated CABG (coronary artery bypass grafting) using MiECC (Minimal extracorporeal circulation system).

ELIGIBILITY:
Inclusion Criteria:

* CABG using MPS® or Cardioplexol ®

Exclusion Criteria:

* use of other colloid solution than Cardioplexol ® or MPS®
* other inventions than CABG
* myocardial infarction <7 days before CABG
* patients denial of data use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing isolated CABG (coronary artery bypass grafting) using MiECC (Minimal extracorporeal circulation system) at the department of cardial surgery University Hospital Basel Switzerland
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2010-02-28 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Change in lab values for cardial biomarkers | perioperative during hospital stay for CABG
  cardial biomarkers measured are high sensitive troponin T (hs-TrT), Creatinkinase, (CK) Creatinkinase myocardial type (CK-MB)

SECONDARY OUTCOMES:
mortality | 30 days after CABG
  death after coronary artery bypass grafting
need for intensive care unit | perioperative during hospital stay for CABG
  duration of stay at intensive care unit
dysrhythmia | perioperative during hospital stay for CABG
  rhythm disturbance after coronary artery bypass grafting
bleeding | perioperative during hospital stay for CABG
  bleeding complication after coronary artery bypass grafting

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Reuthebuch, PD MD, Principal Investigator — University Hospital Basel, CH-4031 Basel
Locations (1):
- Klinik für Herzchirurgie, Universitätsspital Basel, Basel, Switzerland